CLINICAL TRIAL: NCT02014077
Title: VATS( Video-Assisted Thoracoscopy ) Compared to Reinsertion of a Thoracostomy Tube for Persistent Haemothorax A Single Center Prospective Randomized Study
Brief Title: VATS ( Video-Assisted Thoracoscopy) Compared to Reinsertion of a Thoracostomy Tube for Persistent Haemothorax
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cape Town (Other)
Responsible Party: Principal Investigator, Sorin Edu, Dr, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 119/2013
Record Dates: First submitted 2013-12-05; First posted 2013-12-17 (Estimated); Last update posted 2020-01-29 (Actual); Status verified 2020-01

CONDITIONS: Haemothorax; Empyema
Keywords: VATS( Video-Assisted Thoracoscopy ); Thoracostomy Tube; Empyema; Thoracotomy
MeSH Terms: conditions — Hemothorax; Empyema | interventions — Thoracic Surgery, Video-Assisted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Thoracostomy Tube (Active Comparator): patients selected for thoracostomy tube reinsertion after failure of drainage with first thoracostomy tube for traumatic haemothorax
  Interventions: Procedure: Thoracostomy Tube reinsertion
- VATS (Active Comparator): patients selected for VATS after failure of first thoracostomy tube drainage of traumatic haemothorax will undergo a Video-Assisted Thoracoscopic clearance of the persistent/retained haemothorax
  Interventions: Procedure: VATS ( Video-Assisted Thoracoscopy )

INTERVENTIONS:
Procedure: VATS ( Video-Assisted Thoracoscopy ) — the patients were randomized to a Video-Assisted thoracoscopy( VATS )for retained haemothorax
  Arms: VATS
Procedure: Thoracostomy Tube reinsertion — the patient is randomized to reinsertion of a Thoracostomy Tube for retained haemothorax
  Arms: Thoracostomy Tube

SUMMARY:
This is a prospective, randomized study comparing VATS( Video-Assisted Thoracoscopy ) to reinsertion of a Thoracostomy Tube in patients with retained haemothorax. The hypothesis is that early VATS as opposed to reinsertion of a thoracostomy tube , will lead to less complications and shorter hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological diagnosis of retained haemothorax
* Thoracostomy tube blockage or failure to drain

Exclusion Criteria:

* more than one attempt at thoracostomy tube drainage
* unable to consent to trial
* coexisting pathology requiring other interventions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2014-01; Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
duration of hospitalization | patients will be followed during their hospital stay, average 5-14 days
  number of days spent in hospital

SECONDARY OUTCOMES:
number of patients that develop empyema | 2 months form initial injury
  each arm of the study will be monitored for septic complications , specifically empyema of the pleural cavity

OTHER OUTCOMES:
number of patients requiring thoracotomy | 2 months from initial injury
  the patients that develop empyema will require a thoracotomy for clearance of the pleural cavity

CONTACTS AND LOCATIONS:
Overall Officials: Sorin Edu, MD,FCS, Principal Investigator — University of Cape Town
Locations (1):
- Trauma Center, Groote Schuur Hospital,University of Cape Town, Cape Town, Western Cape, South Africa